CLINICAL TRIAL: NCT00714558
Title: Pharmacokinetics of Fentanyl Citrate Following Intravenous (i.v.) and Oral Routes of Administration in Healthy Subjects
Brief Title: Pharmacokinetics of Fentanyl Following Intravenous and Oral Routes of Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR003253
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Biological Availability
Keywords: Pharmacokinetics; Administration, Oral; Naltrexone; Biological Availability; Infusions, Intravenous; Fentanyl; Safety; Naloxone
MeSH Terms: interventions — Fentanyl; Naltrexone; Naloxone

INTERVENTIONS:
Drug: Fentanyl citrate; Naltrexone; Naloxone

SUMMARY:
The purpose of the study is to compare the pharmacokinetics of fentanyl following i.v. and oral administration in healthy volunteers, and to assess the bioavailability of fentanyl following oral administration. Moreover, safety is assessed.

DETAILED DESCRIPTION:
Fentanyl, is an opioid (morphine-like) drug, that has been demonstrated to be an effective pain-killer medication by the i.v. and transdermal (through skin) routes. Fentanyl is used just before, during, and after surgery for its sedative and pain-relieving actions. In addition, fentanyl is currently marketed for transdermal use (Duragesic fentanyl transdermal patch) for the management of chronic pain. The information on the bioavailability of fentanyl solution, following the oral route of administration, is sparse. This is a single-center, randomized (study drug assigned by chance), open-label, 2-treatment, 2-period, crossover study. Healthy volunteers were randomly assigned to 1 of the 2 treatment sequences (AB or BA) with a washout period of 6 to 14 days between treatments. The washout period commenced the day of dosing, after drug administration. Prior to the first treatment period, each healthy volunteer was challenged with naloxone to ensure that he/she was not dependent on morphine-like drugs. A negative naloxone challenge test was required for the healthy volunteer to be eligible for participation in the study. Each healthy volunteer received a 50 mg naltrexone tablet starting 14 hours before dosing and then twice daily ending 24 hours after dosing to block the fentanyl effects. Blood samples were collected, from the arm opposite to the 1 selected for fentanyl i.v administration, for determination of blood fentanyl levels at the scheduled time points. Pulse, blood pressure, breathing rate, body temperature were recorded to monitor the safety. The healthy volunteers were monitored for respiratory depression every 30 minutes during sleep periods. The healthy volunteers remained in the clinic throughout the blood sample collection periods, and were monitored for adverse events throughout the study.

Treatment A: 300 mcg fentanyl citrate administered i.v. over 15 minutes. The 300 mcg (6 mL) i.v. solution was diluted and infused at a rate of 1 mL/minute. Treatment B: 1 mg fentanyl citrate solution administered orally. One mg fentanyl citrate was ingested in 20 mL solution; Naltrexone (50 mg) was administered orally to each healthy volunteer in both periods starting 14 hours before dosing, and twice daily through 24 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non smoker, men and nonpregnant nonlactating women
* Weighing a minimum of 60 kg and were within 15% of ideal weight for height as described in the Metropolitan Life Insurance Height and Weight Standards
* Who did not have a history or show presence of drug or alcohol dependence or abuse
* And who had, after sitting for 5 minutes, blood pressure between the ranges of 100 to 150 mm Hg systolic and 50 to 90 mm Hg diastolic. Any decrease in systolic blood pressure after standing for 2 minutes had to be less than or equal to 20 mm Hg

Exclusion Criteria:

* History of chronic obstructive pulmonary disease or any other lung disease, such as asthma, that would cause carbon dioxide retention
* Known allergy or hypersensitivity to fentanyl or other opioids, naltrexone or naloxone
* Usage of prescription medication (except for birth control medications, sex-hormone replacement or vitamins) within 14 days before Day 1, monoamine oxide inhibitors within 21 days prior to Day 1, over-the-counter medication (except for vitamin supplements or acetaminophen less than 2 gm/day) or herbal medication within 3 days prior to Day 1, alcohol, grapefruit juice, or caffeine within 48 hours before dosing
* Consumption of more than 450 mg of caffeine per day (eg, approximately 5 cups of tea, 3 cups of regular coffee, or 8 cans of cola)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2003-04; Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the pharmacokinetics of fentanyl citrate following i.v. and oral routes of administration in healthy volunteers, and to assess the absolute bioavailability of fentanyl citrate following oral administration.

SECONDARY OUTCOMES:
Assessment of safety. Vital signs, Physical examination, clinical laboratory tests, and electrocardiogram were performed at screening and study termination. Additionally, vital signs were recorded on Days 1 and 2 of both treatment periods.

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — Alza Corporation, DE, USA

REFERENCES:
- See also: Pharmacokinetics of fentanyl following intravenous and oral routes of administration in healthy subjects — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=90&filename=CR003253_CSR.pdf